CLINICAL TRIAL: NCT04333134
Title: A Phase 1, Open-Label, Two-Center Study to Evaluate the Safety and Pharmacokinetics of Single-Dose Fluzoparib in Healthy
Brief Title: A Trial of SHR3162 in Healthy Caucasian Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Atridia Pty Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR3162-I-113
Record Dates: First submitted 2020-04-01; First posted 2020-04-03 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2020-07

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — fluzoparib

STUDY DESIGN:
Intervention Model Description: This study will enroll a single cohort of healthy Caucasian subjects with an approximately one-to-one ratio of male to female subjects
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dose level 1 (Experimental): Will enroll a single cohort of 12 healthy Caucasian subjects with an approximately one-to-one ratio of male to female subjectssubjects can be enrolled and dosed simultaneously.
  Interventions: Drug: SHR3162

INTERVENTIONS:
Drug: SHR3162 — Fluzoparib, also known as SHR3162, is an inhibitor of human PARP
  Other Names: Fluzoparib

SUMMARY:
The purpose of this study is to assess the safety and PK characteristics of a single oral dose of fluzoparib in healthy Caucasian and Chinese subjects

ELIGIBILITY:
Inclusion Criteria:

1. Healthy Caucasian subjects, male and female, 18 to 45 years of age, inclusive, and in good health as determined by past medical history, physical examination, vital signs, electrocardiogram, and laboratory tests;
2. Male body weight ≥50 kg, female body weight ≥45 kg, body mass index (BMI) between ≥18.0 and ≤29.0 kg/m2, inclusive;
3. Female subjects agree not to be pregnant or lactating from beginning of the study screening to 90 days after trial completion:

   * A negative blood and urine pregnancy test for females of childbearing potential at Screening and at Check-in, respectively;
   * Females of reproductive potential are willing and able to employ a highly effective method of birth control/contraception to prevent pregnancy; A highly effective method of contraception is defined as one that results in a low failure rate (ie, less than 1% per year), when used consistently and correctly. Females of non-childbearing potential will not be required to use contraception. Females of non-child bearing potential are defined as permanently sterile (eg, due to hysterectomy) or postmenopausal (defined as at least 12 months following cessation of menses without an alternative medical cause and serum FSH levels >25 IU/L).
4. Males agree to refrain from donating sperm and fathering a child during the study and for at least 90 days after fluzoparib administration; male participants must agree to remain abstinent or must ensure a condom is used for all sexual activity (with a male or female partner) for this same duration.
5. Able and willing to refrain from caffeine or caffeine-containing products, alcohol, fruit juices, and smoking/tobacco products from at least 48 hours prior to Check-In until the end of Safety Follow Up;
6. Able and willing to refrain from eating and drinking poppy seed-containing products and grapefruit-related citrus fruits (eg, Seville oranges, pomelos) within 7 days prior to dosing until after collection of the final PK blood sample (Day 4);
7. Able and willing to refrain from strenuous exercise (heavy lifting, weight training, calisthenics, aerobics) within 7 days prior to dosing until after collection of the final PK blood sample (Day 4);
8. Willing and able to comply with all scheduled visits, study procedures, and provides written informed consent.

Exclusion Criteria:

1. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, neuropsychiatric disease, or any condition that may affect drug absorption, distribution, metabolism, and excretion;
2. Had a severe infection, trauma or major surgery within 4 weeks of screening and at Check-In; plan to have a surgery during the trial;
3. A past medical history of ECG abnormalities, documented cardiac arrhythmias, or cardiovascular disease; or QTcF interval >450 msec for males, >470 msec for females, or <300 msec;
4. Subject's systolic blood pressure (SBP) is >140 or <90 mmHg, diastolic blood pressure (DBP) is >90 or <50 mmHg, resting heart rate <40 or >100 bpm, and respiratory rate <10 or >20 breaths/min at Screening or Check-in after resting in a semi-supine position for 5 minutes. Vitals can be repeated twice (a minimum of 1 to 2 minutes apart) based on the investigator's judgment;
5. History of immunodeficiency including seropositivity for human immunodeficiency virus (HIV), or other acquired or congenital immune-deficient disease, or any active systemic viral infection requiring therapy (eg, hepatitis B or C);
6. Subject has a history of type 1 hypersensitivity to any medication;
7. Subject has evidence of substance abuse, a history of substance abuse, or is positive for drugs of abuse (eg, methamphetamines, opiates, methadone, cocaine, amphetamines, cannabinoids, tricyclic antidepressants, phencyclidine, barbiturates, benzodiazepines), or alcohol at Screening and Check-in (Day -1);
8. History of symptomatic hypoglycemia;
9. Subjects who smoke more than 5 cigarettes per day or will not refrain from smoking starting from at least 48 hours prior to screening and check-in on Day -1, and during the study;
10. History of regular alcohol consumption in the past 3 months exceeding an average weekly intake of 14 standard drinks; 1 drink=5 ounces [150 mL] of wine or 12 ounces [360 mL] of beer or 1.5 ounces [45 mL] of hard liquor;
11. Subject has used prescription medications within 14 days or, as per PI discretion, over-the-counter medications, dietary/nutritional supplements (except hormonal contraceptives, paracetamol under 2 grams/day, vitamin supplements) within 7 days or 5 half-lives prior to fluzoparib administration;
12. Treatment with an investigational drug within 3 months (or 5 half-lives, whichever is longer) of dosing;
13. Use of medications affecting liver metabolism within 1 month of screening;
14. Blood donation or loss of more than 200 mL of blood within 1 month of screening; or blood donation or loss of more than 400 mL of blood within 3 months of screening; or received blood within 8 weeks of screening;
15. Any other major illness/condition that, in the investigator's judgment, substantially increased the risk associated with the subject's participation in and completion of the study or could preclude the evaluation of the subject's response.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2020-04-17 (Actual); Primary Completion 2020-05-15 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic - Cmax | Pre-dose, 0.25, 0.5, 1, 1.5, 2 , 3, 4, 6, 8, 10, 24, 48, and 72 hr post-dose
  Maximum observed plasma concentration (Cmax) of SHR3162
Pharmacokinetic - AUC∞ | Pre-dose, 0.25, 0.5, 1, 1.5, 2 , 3, 4, 6, 8, 10, 24, 48, and 72 hr post-dose
  Area under the concentration-time curve from time 0 to infinity of SHR3162
Pharmacokinetic - Tmax | Pre-dose, 0.25, 0.5, 1, 1.5, 2 , 3, 4, 6, 8, 10, 24, 48, and 72 hr post-dose
  Time to Cmax of SHR3162
Pharmacokinetic - CL/F | Pre-dose, 0.25, 0.5, 1, 1.5, 2 , 3, 4, 6, 8, 10, 24, 48, and 72 hr post-dose
  Apparent clearance of SHR3162
Pharmacokinetic - Vz/F | Pre-dose, 0.25, 0.5, 1, 1.5, 2 , 3, 4, 6, 8, 10, 24, 48, and 72 hr post-dose
  Apparent volume of distribution during terminal phase of SHR3162
Pharmacokinetic - t1/2 | Pre-dose, 0.25, 0.5, 1, 1.5, 2 , 3, 4, 6, 8, 10, 24, 48, and 72 hr post-dose
  Terminal elimination half-life of SHR3162

SECONDARY OUTCOMES:
Adverse events | Screening up to study completion, approximately 5 weeks
  Number of subjects with adverse events (AEs)
Laboratory results | Screening up to study completion, approximately 5 weeks
  Number of subjects with laboratory tests findings of potential clinical importance
Vital signs | Screening up to study completion, approximately 5 weeks
  Incidence of vital sign abnormalities
Electrocardiogram | Screening up to study completion, approximately 5 weeks
  Number of subjects with clinically significant abnormal ECG QT Interval

CONTACTS AND LOCATIONS:
Locations (1):
- Atridia Pty Limited, Sydney, New South Wales, Australia